CLINICAL TRIAL: NCT00660127
Title: The Effect of Visual Stimuli on Itch Perception Intensity in Healthy and Atopic Dermatitis Patients
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 00002112; 32018
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2008-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to assess whether seeing other people itch affects itch perception in patients with atopic dermatitis and healthy subjects.

DETAILED DESCRIPTION:
The objectives of this study are to quantitatively assess the effect of visual stimuli on perception of itch and to assess if visual stimuli affect individuals with atopic dermatitis differently than healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women who are between 18 and 65 years of age
* Diagnosis of moderate to severe atopic dermatitis including involvement of the forearm confirmed by published consensus diagnostic criteria35 (except for healthy control subjects). Severity of AD will be based on an investigator's global assessment score (IGA).
* Subjects must be in general good health with no other skin disease, disease state or physical condition which would impair evaluation of their skin or which would increase their health risk by study participation
* Women of child bearing potential will be required to have a negative pregnancy test in order to enroll in the study and will be required to maintain adequate birth control throughout the study.
* All subjects in Groups 1 and 3 will be required to cease use of oral antihistamines for a period of one week prior to and during the study visit.
* Subjects in Groups 1 and 3 must cease using topical agents on the forearm where experimentation is going to be performed at least 1 week prior. Topical agents can be used in all other parts of the body.
* Baseline COVAS ratings of more than 9/100 after histamine iontophoresis at the screening visit

Exclusion Criteria:

* Adults over age 65
* Children less than 18 years of age
* Unable to complete the required measures
* Currently enrolled in any investigational study in which the subject is receiving any type of drug, biologic, or non-drug therapy and subjects undergoing treatment with another investigational drug or approved therapy for investigational use within 28 days prior to study participation
* Consumption of more than 4 caffeinated beverages per day
* Current treatment with oral lipophilic beta blockers, opioids, glucocorticoids, theophylline, antihistamines or other medications known to interfere with itch perception or heart rate variability as determined by the investigators
* Uncontrolled asthma or COPD
* Uncontrolled thyroid disease
* Poorly controlled diabetes mellitus
* Poorly compensated congestive heart failure
* Use of illicit drugs
* History of chronic urticaria
* History of anaphylactic shock
* History of neuropathy causing disease such as diabetes and uremia
* Allergy to histamine
* Blindness
* Baseline COVAS ratings of less than 9/100 after histamine iontophoresis at the screening visit
* Subject participation in more than one group.
* Positive pregnancy test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: general community population
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gil Yosipovitch, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States